CLINICAL TRIAL: NCT02123823
Title: A Phase Ib/II Randomized Study of BI 836845 in Combination With Exemestane and Everolimus Versus Exemestane and Everolimus Alone in Women With Locally Advanced or Metastatic Breast Cancer
Brief Title: BI 836845 in Estrogen Receptor Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1280.4; 2013-001110-15 (EudraCT Number)
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Everolimus; exemestane; xentuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- everolimus 10 mg + exemestane 25 mg - Phase II (Active Comparator): Subjects received a single oral dose once daily (qd) of 2x 5 mg (10 mg total) tablets of everolimus and 1 tablet of 25 mg exemestane starting on Day 1 continously until disease progression, intolerable AEs or other reason necessitating withdrawal.
  Interventions: Drug: Everolimus; Drug: Exemestane
- xentuzumab (BI 836845) 1000 mg + everolimus 10 mg + exemestane 25 mg - Phase II (Experimental): Subjects received a single dose of 1000 milligram (mg) BI 836845 (xentuzumab) as a 1 hour (h) intravenous infusion once a week on Day 1, 8, 15 and 22 in a 28-day course until disease progression, intolerable AEs or other reason necessitating withdrawal. Subjects also received a single oral dose once daily (qd) of 2x 5 mg (10 mg total) tablets of everolimus and 1 tablet of 25 mg exemestane starting on Day 1 continously until disease progression, intolerable AEs or other reason necessitating withdrawal. Administration of xentuzumab was stopped after 28th October 2016, and participants in this group who remained in the trial could continue with everolimus 10 mg + exemestane 25 mg.
  Interventions: Drug: Everolimus; Drug: Exemestane; Drug: BI 836845
- xentuzumab (BI 836845) 750 mg + everolimus 10 mg + exemestane 25 mg - Phase Ib (Experimental): Subjects received a single dose of 750 milligram (mg) BI 836845 (xentuzumab) as a 1 hour (h) intravenous infusion once a week on Day 1, 8, 15 and 22 in a 28- day course until disease progression, intolerable AEs or other reason necessitating withdrawal. Subjects also received a single oral dose once daily (qd) of 2x 5 mg (10 mg total) tablets of everolimus and 1 tablet of 25 mg exemestane starting 7 days before first administration of BI 836845 (xentuzumab) continously until disease progression, intolerable AEs or other reason necessitating withdrawal.
  Interventions: Drug: Everolimus; Drug: Exemestane; Drug: BI 836845
- xentuzumab (BI 836845) 1000 mg + everolimus 10 mg + exemestane 25 mg - Phase Ib (Experimental): Subjects received a single dose of 1000 milligram (mg) BI 836845 (xentuzumab) as a 1 hour (h) intravenous infusion once a week on Day 1, 8, 15 and 22 in a 28-day course until disease progression, intolerable AEs or other reason necessitating withdrawal. Subjects also received a single oral dose once daily (qd) of 2x 5 mg (10 mg total) tablets of everolimus and 1 tablet of 25 mg exemestane starting 7 days before first administration of BI 836845 (xentuzumab) continously until disease progression, intolerable AEs or other reason necessitating withdrawal.
  Interventions: Drug: Everolimus; Drug: Exemestane; Drug: BI 836845

INTERVENTIONS:
Drug: Everolimus — 10mg dose
Drug: Exemestane — Fixed dose at 25mg
Drug: BI 836845 — 1000 mg, recommended dose per Phase Ib part. Human monoclonal antibody. Dose escalation in Phase Ib. 2 dose levels (high or low) depending on the dose cohort explored
  Other Names: xentuzumab
  Arms: xentuzumab (BI 836845) 1000 mg + everolimus 10 mg + exemestane 25 mg - Phase II; xentuzumab (BI 836845) 1000 mg + everolimus 10 mg + exemestane 25 mg - Phase Ib; xentuzumab (BI 836845) 750 mg + everolimus 10 mg + exemestane 25 mg - Phase Ib

SUMMARY:
Phase Ib / II study to determine the Maximum Tolerated Dose and Recommended Phase II Dose, and to evaluate the safety and antitumour activity, of BI 836845 and everolimus in combination with exemestane in women with HR+/HER2- advanced breast cancer

ELIGIBILITY:
Inclusion criteria:

* Histologically-confirmed locally advanced (aBC) or metastatic breast cancer (mBC) not deemed amenable to curative surgery or curative radiation therapy
* Tumors are positive for estrogen-receptor (ER) and/or progesterone receptor (PgR).
* Tumors must be negative for HER2 per local lab testing.
* Must have adequate archival tumor tissue from surgery or biopsy.
* Postmenopausal female patients aged >=18 years old.
* Objective evidence of recurrence or progressive disease on or after the last line of systemic therapy for breast cancer prior to study entry
* The patient is disease refractory to non-steroidal aromatase inhibitor (letrozole and/or anastrozole)
* Patients must have: a) Measurable lesion according to RECIST version 1.1 (R09-0262) or b) Bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable lesion as defined above
* Eastern Cooperative Oncology Group performance score <= 2.
* Life expectancy of >= 6 months in the opinion of the investigator
* Fasting plasma glucose < 8.9 mmol/L (< 160 mg/dL) and HbA1c < 8.0%
* Adequate organ function
* Recovered from any previous therapy related toxicity to <= Grade 1 at study entry (except for stable sensory neuropathy <=Grade 2 and alopecia)
* Written informed consent that is consistent with ICH-GCP guidelines and local regulations

Inclusion criteria for the biopsy substudy are identical to the main study of the phase II part except for the following two inclusion criteria:

* Fresh tumor biopsy should be taken when deemed safe and feasible by the investigator and upon informed consent by the patient. Bone lesion is not recommended for biopsy
* Patients eligible to undergo tumor biopsy should have normal coagulation parameters (INR and PTT within normal range)

Exclusion criteria:

* Previous treatment with agents targeting on IGF pathway, phosphoinositide 3-kinase (PI3K) signaling pathway, protein kinase B (AKT), or mammalian target of rapamycin (mTOR) pathways
* Prior treatment with exemestane (except adjuvant exemestane stopped >12 months prior to start of study treatment as long as the patient did not recur during or within 12 months after the end of adjuvant exemestane)
* Known hypersensitivity to monoclonal antibody, mTOR inhibitors (e.g. sirolimus), or to the excipients of any study drugs
* Ovarian suppression by ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist
* Less than one week after receiving immunization with attenuated live vaccines prior to study treatment
* Radiotherapy within 4 weeks prior to the start of the study treatment, except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within two weeks prior to study treatment
* Chemotherapy, biological therapy (other than bevacizumab), immunotherapy or investigational agents within 5 half-life of the drug or within two weeks prior to the start of study treatment, whichever is longer; bevacizumab treatment within 4 weeks prior to start of study treatment (this criterion concerns anti-cancer therapy only)
* Hormonal treatment for breast cancer within 2 weeks prior to start of study treatment
* Major surgery in the judgement of the investigator within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use except Topical applications, inhaled sprays, eye drops or local injections or Patients on stable low dose of corticosteroids for at least two weeks before study entry
* Chronic hepatitis B infection, chronic hepatitis C infection and/or known HIV carrier
* QTcF prolongation > 470 ms or QT prolongation deemed clinically relevant by the investigator
* Disease that is considered by the investigator to be rapidly progressing or life threatening such as extensive symptomatic visceral disease including hepatic involvement and pulmonary lymphangitic spread of tumor
* History or current presence of brain or other CNS metastases
* Bilateral diffuse lymphangitic carcinomatosis (in lung)
* Hypokalemia of Grade >1
* History of another primary malignancy within 5 years, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer
* Family history of long QT syndrome
* Any concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety and anti-tumor activity of the test drug(s)
* Patients being treated with drugs recognized being strong or moderate CYP3A4 and/or PgP inhibitors and/or strong CYP3A4 inducers within 2 weeks prior to study entry
* Patients received more than two lines of chemotherapy for locally advanced or metastatic breast cancer (For the Phase II: more than one line)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (38):
- Austria (2):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Wilhelminenspital, Vienna
- Belgium (8):
  - Brussels - UNIV UZ Brussel, Brussels
  - Brussels - UNIV Saint-Luc, Brussels
  - Charleroi - HOSP Grand Hôpital de Charleroi, Charleroi
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Liège - HOSP St-Joseph, Liège
  - CHU UCL Namur - Site De Sainte-Elisabeth, Namur
- France (6):
  - HOP Jean Minjoz, Besançon
  - INS Paoli-Calmettes, Marseille
  - CTR Catherine de Sienne, Nantes
  - HOP Européen G. Pompidou, Paris
  - INS Curie, Paris
  - Ctr Cario, Plerin Sur Mer
- St. Vincent's University Hospital, Dublin, Ireland
- Maastricht University, Maastricht, Netherlands
- South Korea (3):
  - National Cancer Center, Goyang
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (9):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico de Valencia, Valencia
- Centrummottagningen, Stockholm, Sweden
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Ninewells Hospital & Medical School, Dundee
  - St Bartholomew's Hospital, London
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Dercle L, McGale J, Zhao B, Schmitt J, Peltzer A, Schwartz LH, Amend M. Artificial intelligence and radiomics biomarkers for treatment response prediction in advanced HER2-negative breast cancer. Breast. 2025 Dec;84:104571. doi: 10.1016/j.breast.2025.104571. Epub 2025 Sep 3. PMID 40974664
- [Derived] Schmid P, Sablin MP, Bergh J, Im SA, Lu YS, Martinez N, Neven P, Lee KS, Morales S, Perez-Fidalgo JA, Adamson D, Goncalves A, Prat A, Jerusalem G, Schlieker L, Espadero RM, Bogenrieder T, Huang DC, Crown J, Cortes J. A phase Ib/II study of xentuzumab, an IGF-neutralising antibody, combined with exemestane and everolimus in hormone receptor-positive, HER2-negative locally advanced/metastatic breast cancer. Breast Cancer Res. 2021 Jan 15;23(1):8. doi: 10.1186/s13058-020-01382-8. PMID 33451345
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a phase Ib/II, randomized, open label study to determine the maximum tolerated dose (MTD) and the recommended phase II dose and to evaluate the anti-tumor activity of BI 836845 (xentuzumab) in combination with exemestane and everolimus versus exemestane and everolimus alone in women with locally advanced or metastatic breast cancer.
Pre-assignment Details: Only subjects that met all inclusion + none of exclusion criteria were to be entered. Subjects were free to withdraw from clinical trial at any time for any reason given. If subject continued to take trial drug, close monitoring was adhered to + adverse events recorded. Rules were implemented in all trials whereby doses would be reduced if required. If further events were reported, subject would be withdrawn from trial. Symptomatic treatment of tumor associated symptoms were allowed throughout.
Groups:
- Xentuzumab (BI 836845) 750 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib: Subjects received a single dose of 750 milligram (mg) BI 836845 (xentuzumab) as a 1 hour (h) intravenous infusion once a week on Day 1, 8, 15 and 22 in a 28-day course until disease progression, intolerable AEs or other reason necessitating withdrawal.
  Subjects also received a single oral dose once daily (qd) of 2x 5 mg (10 mg total) tablets of everolimus and 1 tablet of 25 mg exemestane starting 7 days before first administration of BI 836845 (xentuzumab) continously until disease progression, intolerable AEs or other reason necessitating withdrawal.
Period: Overall Study
Arm/Group | Xentuzumab (BI 836845) 750 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Started (randomized) | 3 | 21 | 70 | 70
Treated | 3 | 21 | 70 | 69
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 21 | 70 | 70
Not completed — Lack of Efficacy | 0 | 2 | 8 | 10
Not completed — Progressive disease | 3 | 19 | 52 | 53
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 2
Not completed — Adverse Event | 0 | 0 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Treated set (Phase Ib only): This patient set included all patients who were documented to have received and taken at least one dose of any study medication during the treatment cycles (from Day 1).
  Randomised set (RS) (Phase II only): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with exemestane and everolimus or exemestane and everolimus alone as randomised.
Groups:
- Total: Total of all reporting groups
Arm/Group | Xentuzumab (BI 836845) 750 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II | Total
Number analyzed (Participants) | 3 | 21 | 70 | 70 | 164
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.00 (8.00) | 64.33 (7.84) | 60.17 (9.61) | 60.67 (9.07) | 60.90 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 21 | 70 | 70 | 164
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 5 | 8
  Not Hispanic or Latino | 3 | 19 | 62 | 57 | 141
  Unknown or Not Reported | 0 | 0 | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 21 | 53 | 51 | 128
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) - Phase II Part
Description: Progression-free survival (PFS) in the phase II part is presented. Progression-free survival (PFS) was defined as the time from randomisation until radiological tumour progression according to RECIST 1.1, or death from any cause, whichever occurred earlier. Clinical disease progression was not considered for determination of a PFS event, unless the outcome of the progression was death. The cut-off date was 25th November 2016. At cut-off date, xentuzumab was discontinued in all patients in the experimental arm per sponsor decision, recruitment was also terminated. Patients who discontinued xentuzumab treatment continued with everolimus 10 mg + exemestane 25 mg treatment.
Time Frame: From randomisation until radiological tumour progression according to RECIST 1.1, or death from any cause or data cut-off (25Nov2016), up to 30 months.
Population: Randomised set (RS): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab (BI 836845) in combination with exemestane and everolimus or exemestane and everolimus alone as randomised.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Number analyzed (Participants) | 70 | 70
Months | 7.3 [3.3 to NA] — Not enough events to calculate the value | 5.6 [3.7 to 9.1]
Statistical Analysis 1: Comparison: Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II vs Everolimus 10 mg + Exemestane 25 mg - Phase II; Test type: Other; p = 0.9057, Log Rank; Two-sided log-rank test stratified for visceral involvement; Hazard Ratio, log = 0.97, 95% CI 2-sided [0.57 to 1.65] — Cox proportional hazards model stratified for visceral involvement

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) - Phase Ib Part
Description: Number of patients with dose limiting toxicity (DLT) in phase Ib part is presented.
Time Frame: From first administration of study treatment until end of first treatment cycle, up to 28 days.
Population: Maximum tolerated dose (MTD) set: The MTD set defined the set of patients in the Phase Ib part who were fully evaluable for determination of the MTD in the first treatment course. Patients in the TS who were replaced within the MTD evaluation period in the first part of the trial were excluded from the determination of the MTD.
Measure: Count of Participants; unit: Participants
Arm/Group | Xentuzumab (BI 836845) 750 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1

3. Primary Outcome: Maximum Tolerated Dose (MTD) - Phase Ib Part
Description: The Maximum Tolerated Dose (MTD) in this study was defined as the highest dose level examined of trial medication, at which no more than 1 out of 6 patients experienced a DLT during the MTD evaluation period.
  The MTD evaluation period was defined as the time from the first administration of xentuzumab up to start of cycle 2.
  A "3+3" Phase Ib dose finding phase was performed to determine the MTD.
Time Frame: up to 28 days.
Population: as for outcome 2
Measure: Number; unit: milligrams (mg)
Groups:
- Xentuzumab (BI 836845): Treatment group "xentuzumab (BI 836845) comprises all dose cohorts during the dose finding phase, that is, "xentuzumab (BI 836845) 750 mg + everolimus 10 mg + exemestane 25 mg" and "xentuzumab (BI 836845) 1000 mg + everolimus 10 mg + exemestane 25 mg".
  All patients were administered doses of xentuzumab (BI 836845) as a 1 hour (h) intravenous infusion once a week on Day 1, 8, 15 and 22 in a 28-day course in the absence of disease progression, intolerable AEs or other reason necessitating withdrawal.
  Subjects also received a single oral dose once daily (qd) of 2x 5 mg (10 mg total) tablets of everolimus and 1 tablet of 25 mg exemestane starting 7 days before first administration of BI 836845 (xentuzumab) continously in the absence of disease progression, intolerable AEs or other reason necessitating withdrawal.
Arm/Group | Xentuzumab (BI 836845)
Number analyzed (Participants) | 9
milligrams (mg) | 1000

4. Secondary Outcome: Number of Patients With Objective Response (OR) - Phase II Part
Description: Objective response (OR) - phase II part is presented. Objective response (OR), defined as best overall response of complete response (CR) or partial response (PR), where best overall response was determined according to RECIST 1.1 from date of randomisation until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.
Time Frame: From randomisation until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy or data cut-off (25Nov2016), up to 30 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Number analyzed (Participants) | 70 | 70
Participants | 5 [2.4 to 15.9] | 7 [4.1 to 19.5]
Statistical Analysis 1: Comparison: Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II vs Everolimus 10 mg + Exemestane 25 mg - Phase II; Test type: Other; p = 0.5598, Regression, Logistic; Odds ratio and p-value are obtained from logistic regression model adjusted for visceral involvement at screening; Odds Ratio, log = 0.70, 95% CI 2-sided [0.20 to 2.32] — An odds ratio >1 indicates a benefit to the xentuzumab arm

5. Secondary Outcome: Time to Progression (TTP) - Phase II Part
Description: Time to progression (TTP) is presented. Time to progression (TTP), defined as the time from the date of randomization until the date of the first objective tumour progression according to RECIST 1.1.
Time Frame: From randomisation until the date of the first objective tumour progression according to RECIST 1.1. or data cut-off (25Nov2016), up to 30 months.
Population: Randomised set (RS): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab (BI 836845) in combination with exemestane and everolimus or exemestane and everolimus alone as randomised. Only patients with progression were analysed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Number analyzed (Participants) | 70 | 70
Months | 7.3 [3.7 to NA] — Not enough events to calculate the value | 5.6 [5.3 to 9.1]
Statistical Analysis 1: Comparison: Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II vs Everolimus 10 mg + Exemestane 25 mg - Phase II; Test type: Other; p = 0.9146, Log Rank; Two-sided log-rank test stratified for visceral involvement; Hazard Ratio, log = 1.03, 95% CI 2-sided [0.59 to 1.80] — Cox proportional hazards model stratified for visceral involvement

6. Secondary Outcome: Number of Patients With Disease Control (DC) - Phase II Part
Description: Disease control is defined as best overall response of complete response (CR) or partial response (PR), or stable disease (SD) >= 24 weeks, or Non-CR/Non-PD for >= 24 weeks. PD=Progressive disease.
Time Frame: From randomisation until data cut-off (25Nov2016), up to 30 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Number analyzed (Participants) | 70 | 70
Participants | 13 [10.3 to 29.7] | 17 [14.8 to 36.0]
Statistical Analysis 1: Comparison: Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II vs Everolimus 10 mg + Exemestane 25 mg - Phase II; Test type: Other; p = 0.4008, Regression, Logistic; Odds ratio and p-value are obtained from logistic regression model adjusted for visceral involvement; Odds Ratio, log = 0.70, 95% CI 2-sided [0.31 to 1.59] — An odds ratio >1 indicates a benefit to the xentuzumab arm

7. Secondary Outcome: Time to Objective Response - Phase II Part
Description: Time to objective response is presented. Time to objective response is defined as the time from randomisation until first documented complete response (CR) or partial response (PR).
Time Frame: From randomisation until first documented complete response (CR) or partial response (PR) or data cut-off (25Nov2016), up to 30 months.
Population: Randomised set (RS): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab (BI 836845) in combination with exemestane and everolimus or exemestane and everolimus alone as randomised. Only patients with objective response were analysed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Number analyzed (Participants) | 5 | 7
Months | 3.7 [3.6 to 5.3] | 1.8 [1.7 to 5.3]

8. Secondary Outcome: Duration of Objective Response - Phase II Part
Description: Duration of objective response is presented. Duration of objective response is defined as the time from first documented complete response (CR) or partial response (PR) until the earliest of disease progression or death among patients with objective response (OR).
Time Frame: From randomisation until the earliest of disease progression or death or data cut-off (25Nov2016), up to 30 months.
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Number analyzed (Participants) | 5 | 7
Months | 5.6 [5.6 to 5.6] | NA [NA to NA] — Not enough events to calculate the value

9. Secondary Outcome: Duration of Disease Control - Phase II Part
Description: Duration of disease control is presented. Duration of disease control is defined as the time from randomisation until the earliest of disease progression or death, among patients with disease control.
Time Frame: From randomisation until the earliest of disease progression or death or data cut-off (25Nov2016), up to 30 months.
Population: Randomised set (RS): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab (BI 836845) in combination with exemestane and everolimus or exemestane and everolimus alone as randomised. Only patients with disease control were analysed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
Number analyzed (Participants) | 13 | 17
Months | NA [10.9 to NA] — Not enough events to calculate the value | 9.3 [9.1 to NA] — Not enough events to calculate the value

ADVERSE EVENTS:
Time Frame: For all AEs including all-cause mortality: Phase Ib: from first dose until last dose + 42 days of residual effect period, up to 54.3 months + 42 days Phase II: from first dose until last dose + 42 days of residual effect period, up to 37.7 months + 42 days
Description: Treated set (Phase Ib): including all patients who were documented to have received and taken at least one dose of any study medication during the treatment cycles (from Day 1).
  Randomised set (Phase II): including all randomised patients, regardless of whether or not they received treatment. Patients were assigned to xentuzumab + exemestane (Ex) + everolimus (Ev) or Ex+Ev as randomised.
  Adverse events were reported by initial treatment groups as planned in the Statistical Analysis Plan.
Arm/Group | Xentuzumab (BI 836845) 750 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II | Everolimus 10 mg + Exemestane 25 mg - Phase II
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/21 | 9/70 | 11/69
Serious Adverse Events (participants affected / at risk) | 3/3 | 10/21 | 20/70 | 29/69
Other Adverse Events (participants affected / at risk) | 3/3 | 21/21 | 70/70 | 68/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xentuzumab (BI 836845) 750 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib (N=3) | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib (N=21) | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II (N=70) | Everolimus 10 mg + Exemestane 25 mg - Phase II (N=69)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Scrub typhus (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Reexpansion pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 3
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xentuzumab (BI 836845) 750 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib (N=3) | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase Ib (N=21) | Xentuzumab (BI 836845) 1000 mg + Everolimus 10 mg + Exemestane 25 mg - Phase II (N=70) | Everolimus 10 mg + Exemestane 25 mg - Phase II (N=69)
Anaemia (Blood and lymphatic system disorders) | 3 | 13 | 16 | 16
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 6 | 7 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 1 | 8 | 20 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 17 | 10
Visual acuity reduced (Eye disorders) | 1 | 0 | 1 | 0
Xerophthalmia (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 11 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 6 | 6
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 3 | 15 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 12 | 31 | 23
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 5 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 3 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 3 | 12
Nausea (Gastrointestinal disorders) | 1 | 9 | 24 | 16
Odynophagia (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 8 | 24 | 26
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 7 | 14 | 15
Asthenia (General disorders) | 3 | 9 | 23 | 24
Calcinosis (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 5 | 6
Fatigue (General disorders) | 0 | 9 | 19 | 17
Influenza like illness (General disorders) | 0 | 0 | 1 | 5
Mucosal dryness (General disorders) | 0 | 2 | 2 | 1
Mucosal inflammation (General disorders) | 3 | 10 | 27 | 22
Oedema peripheral (General disorders) | 1 | 5 | 11 | 16
Pyrexia (General disorders) | 1 | 7 | 10 | 7
Bronchitis (Infections and infestations) | 0 | 1 | 4 | 3
Cystitis (Infections and infestations) | 0 | 2 | 4 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 2 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 5 | 12 | 12
Oral herpes (Infections and infestations) | 0 | 1 | 2 | 4
Paronychia (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 2 | 2 | 3
Tooth abscess (Infections and infestations) | 0 | 2 | 2 | 1
Tooth infection (Infections and infestations) | 0 | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 5 | 10
Urinary tract infection (Infections and infestations) | 0 | 6 | 7 | 9
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 5 | 18 | 11
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 14 | 14
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 1 | 2
Blood cholesterol increased (Investigations) | 0 | 3 | 1 | 6
Blood creatine phosphokinase increased (Investigations) | 2 | 7 | 11 | 7
Blood creatinine increased (Investigations) | 1 | 5 | 3 | 4
Blood glucose increased (Investigations) | 0 | 2 | 1 | 1
Blood iron decreased (Investigations) | 0 | 2 | 1 | 2
Blood phosphorus decreased (Investigations) | 0 | 2 | 3 | 2
Blood triglycerides increased (Investigations) | 1 | 2 | 5 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 5 | 8 | 7
Haemoglobin decreased (Investigations) | 0 | 4 | 2 | 1
Low density lipoprotein increased (Investigations) | 0 | 3 | 3 | 1
Neutrophil count decreased (Investigations) | 1 | 4 | 8 | 2
Platelet count decreased (Investigations) | 2 | 4 | 14 | 3
Weight decreased (Investigations) | 1 | 11 | 6 | 9
Decreased appetite (Metabolism and nutrition disorders) | 1 | 13 | 18 | 22
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 5 | 7 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 11 | 18 | 17
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 5 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 7 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 4 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 7 | 11 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 11 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 12 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 8 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 8 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 8 | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 4 | 5
Dysgeusia (Nervous system disorders) | 1 | 8 | 10 | 9
Headache (Nervous system disorders) | 0 | 5 | 17 | 10
Insomnia (Psychiatric disorders) | 0 | 3 | 8 | 8
Sleep disorder (Psychiatric disorders) | 0 | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 4 | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 0 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 4 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 25 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 12 | 18
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 13 | 12
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 7 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 8 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 5 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 5 | 2 | 4
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6 | 14 | 15
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 25 | 23
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0
Hot flush (Vascular disorders) | 0 | 3 | 4 | 1
Hypertension (Vascular disorders) | 0 | 9 | 8 | 7
Lymphoedema (Vascular disorders) | 0 | 1 | 7 | 2

LIMITATIONS AND CAVEATS:
Xentuzumab was stopped in all patients in the experimental arm per sponsor decision on 28 October 2016 with the implementation of protocol Amendment 3; these patients could continue receiving everolimus plus exemestane. All patients in the experimental arm were to attend for an end of xentuzumab visit (EoXV) after this communication. The EoXV had the same procedures as the end of trial visit (EOTV). Further recruitment was stopped but trial was completed per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT02123823/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT02123823/SAP_001.pdf